CLINICAL TRIAL: NCT03722004
Title: Intestinal and Humoral Immunity of Monovalent Oral Poliovirus Vaccine Type 1 When Administered With and Without Fractional Inactivated Poliovirus Vaccine
Brief Title: Monovalent Oral Poliovirus Vaccine Type 1 Intestinal and Humoral Immunity Study
Acronym: mOPV1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR-18045
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis
Keywords: monovalent oral poliovirus vaccine type 1; bivalent oral poliovirus vaccine; inactivated poliovirus vaccine; fractional inactivated poliovirus vaccine; humoral immunity; intestinal immunity; Bangladesh
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mOPV1 + fIPV 6 weeks (Active Comparator): mOPV1 administered at 6, 10, and 14 weeks and fIPV at 6 weeks.
  Interventions: Biological: mOPV1; Biological: fIPV
- mOPV1 + fIPV 10 weeks (Active Comparator): mOPV1 administered at 6, 10, and 14 weeks and fIPV at10 weeks.
  Interventions: Biological: mOPV1; Biological: fIPV
- mOPV1 only (Active Comparator): mOPV1 administered at 6, 10, and 14 weeks.
  Interventions: Biological: mOPV1
- bOPV only (Active Comparator): bOPV administered at 6, 10, and 14 weeks.
  Interventions: Biological: bOPV

INTERVENTIONS:
Biological: mOPV1 — Monovalent oral poliovirus vaccine type 1 is a type-specific, live, attenuated oral poliovirus vaccine that protects against poliovirus type 1.
  Arms: mOPV1 + fIPV 10 weeks; mOPV1 + fIPV 6 weeks; mOPV1 only
Biological: bOPV — Bivalent oral poliovirus vaccine is a live, attenuated oral poliovirus vaccine that protects against poliovirus types 1 and 3.
  Arms: bOPV only
Biological: fIPV — Fractional dose of inactivated poliovirus vaccine that protects against types 1, 2, and 3 (all polio serotypes). Given as a 0.1 milliliter (mL) dose (fractional) by intradermal injection in lieu of the full 0.5mL dose that is given intramuscularly.
  Arms: mOPV1 + fIPV 10 weeks; mOPV1 + fIPV 6 weeks

SUMMARY:
This is an open-label phase IV randomized clinical trial that will assess intestinal and humoral immunity among infants who receive a combination of monovalent oral poliovirus vaccine type 1 and fractional dose of inactivated poliovirus vaccine, monovalent oral poliovirus vaccine type 1 only, and bivalent oral poliovirus vaccine only.

DETAILED DESCRIPTION:
The risk for circulating vaccine-derived poliovirus (cVDPV) will increase in the years immediately after the cessation of oral poliovirus vaccine (OPV) use in routine immunization programs. Judicious use of type-specific monovalent OPV (mOPV) will be necessary for outbreak response to prevent further paralytic infections and transmission; however, data on the intestinal and humoral immunity induced by mOPV1 are very limited. Furthermore, the additional benefit of fractional dose inactivated poliovirus vaccine (fIPV) on type 1 immunity when given with mOPV1 is unclear. Data on intestinal and humoral immunity of mOPV type 1 (mOPV1) and combination use of mOPV1 and fractional dose of IPV (fIPV) are urgently needed and would be used to inform guidelines for type 1 outbreak response in a post-OPV world. In the immediate future, a strategy of shifting from bivalent OPV (bOPV) to mOPV1 as part of supplemental immunization activities in endemic countries is under consideration but data on intestinal and humoral immunity to support this change does not exist. This trial is designed to address both areas in which data are lacking.

Healthy infants 5 weeks of age will be enrolled at two study clinics in Dhaka, Bangladesh, and randomized to one of four study arms: mOPV1 + fIPV at 6 weeks, mOPV1 + fIPV at 14 weeks, mOPV1 only, and bOPV only. Infants will be followed-up until 18 weeks of age by clinic and household visits. Blood and stool specimens will be collected to test for vaccine response (humoral immunity) and vaccine virus shedding (intestinal immunity).

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 5 weeks of age (range: 35-41 days).
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of fIPV or collection of blood by venipuncture.
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Infection or illness at the enrolment visit (i.e., 5 weeks of age) that a study medical officer judges would prevent the start of study activities at 6 weeks of age (i.e., blood collection and vaccination).
* Receipt of any polio vaccine (OPV or IPV/fIPV) before enrolment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine, or its contents.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).

Ages: 35 Days to 41 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1256 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Vaccine response | Measured four weeks after administration of study vaccine(s). Vaccine response will be measured at 10 weeks, 14 weeks, and 18 weeks of age after 1, 2, and 3 doses of OPV, respectively.
  Dichotomous (yes/no) variable defined as participants who are either seronegative (<1:8 titers) at baseline who become seropositive (≥1:8) after vaccination (seroconversion) or participants who demonstrate a four-fold rise in titers after vaccination between two specimens, e.g. a change from 1:8 to 1:32, after adjusting for expected decay in maternal antibodies. Antibody titers at 6 weeks of age will be the starting point for the expected decline in maternal antibodies, assuming at half-life of 28 days.
Vaccine virus particles | Measured 7 and 14 days after administration of the study vaccine. For Arms B, C, and D, this will be after administration of the first mOPV1 or bOPV dose. For Arms A, B, and C, this will be after the mOPV1 challenge dose at 14 weeks of age.
  Presence or absence of vaccine virus particles in stool specimens.

SECONDARY OUTCOMES:
Reciprocal antibody titers | Measured four weeks after administration of study vaccine(s). Vaccine response will be measured at 10 weeks, 14 weeks, and 18 weeks of age after 1, 2, and 3 doses of OPV, respectively.
  Variable of the observed reciprocal antibody titer results.

CONTACTS AND LOCATIONS:
Locations (1):
- icddr,b study clinics (Mirpur and CTU Dhaka), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snider CJ, Zaman K, Wilkinson AL, Binte Aziz A, Yunus M, Haque W, Jones KAV, Wei L, Estivariz CF, Konopka-Anstadt JL, Mainou BA, Patel JC, Lickness JS, Pallansch MA, Wassilak SGF, Steven Oberste M, Anand A. Poliovirus type 1 systemic humoral and intestinal mucosal immunity induced by monovalent oral poliovirus vaccine, fractional inactivated poliovirus vaccine, and bivalent oral poliovirus vaccine: A randomized controlled trial. Vaccine. 2023 Sep 22;41(41):6083-6092. doi: 10.1016/j.vaccine.2023.08.055. Epub 2023 Aug 29. PMID 37652822